CLINICAL TRIAL: NCT00522353
Title: Effect of Oligofructose Versus Placebo on Body Weight and Satiety Hormone Secretion in Overweight and Obese Adults.
Brief Title: Prebiotic Fiber as a Modifier of Satiety Hormones and Body Weight in Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Raylene Reimer, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UC 20085
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Obesity
Keywords: obesity; weight loss; satiety hormones; body composition; appetite ratings
MeSH Terms: conditions — Obesity; Weight Loss | interventions — oligofructose; fructooligosaccharide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Oligofructose
  Interventions: Dietary Supplement: Oligofructose
- 2 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oligofructose — 21 grams per day in distributed over 3 doses per day for 3 months
  Other Names: Raftilose P95
  Arms: 1
Dietary Supplement: Placebo — 7.89 grams of placebo maltodextrin divided into 3 equal doses per day for 3 months
  Other Names: Maltrin M100
  Arms: 2

SUMMARY:
The purpose of this study is to determine if oligofructose supplementation promotes weight loss in overweight and obese adults.

DETAILED DESCRIPTION:
Obesity is a primary health concern for many western countries as it is linked to several chronic diseases as well as, large health care costs. Although obesity is a multifactorial disease, it is known that levels of satiety hormones including glucagon like peptide-1 (GLP-1) and peptide YY (PYY) are reduced in obesity. The ability of prebiotic fiber to promote weight loss through the production of satiety hormones has been tested previously using rodents. Here it was found that prebiotic supplementation resulted in a decreased energy intake, higher GLP-1 levels in the plasma and increased proglucagon mRNA levels in the gut. This study will address the important question of whether prebiotic fiber supplementation is effective in reducing body weight in overweight or obese human subjects.

ELIGIBILITY:
Inclusion Criteria:

* overweight or class I obese individuals with BMI between 25 kg/m2 and 34.9 kg/m2
* stable body weight in previous 3 months

Exclusion Criteria:

* Type 1 and Type 2 diabetes
* clinically significant cardiovascular abnormalities
* liver or pancreas disease
* major gastrointestinal surgeries
* are pregnant or lactating
* exhibit alcohol or drug dependence
* on drugs influencing appetite
* are following a diet or exercise regime designed for weight loss
* have a body mass greater than 350lb
* chronic use of antacids or bulk laxatives

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-01; Primary Completion 2007-05 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Body weight | 3 months

SECONDARY OUTCOMES:
Plasma satiety hormones | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Raylene A. Reimer, PhD, RD, Principal Investigator — University of Calgary
Locations (1):
- Faculty of Kinesiology, Roger Jackson Centre for Health and Wellness Research, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Parnell JA, Klancic T, Reimer RA. Oligofructose decreases serum lipopolysaccharide and plasminogen activator inhibitor-1 in adults with overweight/obesity. Obesity (Silver Spring). 2017 Mar;25(3):510-513. doi: 10.1002/oby.21763. PMID 28229548
- [Derived] Parnell JA, Reimer RA. Weight loss during oligofructose supplementation is associated with decreased ghrelin and increased peptide YY in overweight and obese adults. Am J Clin Nutr. 2009 Jun;89(6):1751-9. doi: 10.3945/ajcn.2009.27465. Epub 2009 Apr 22. PMID 19386741